CLINICAL TRIAL: NCT00084604
Title: A Multicenter, Open-Label, Phase II Study of Irinotecan, Cisplatin, and Bevacizumab in Patients With Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Irinotecan, Cisplatin, and Bevacizumab in Treating Patients With Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01450; 04-021; NCI-6447; MSKCC-04021; CDR0000365463; N01CM17105 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Bevacizumab; Cisplatin

ARMS (1):
- Treatment (bevacizumab, cisplatin, irinotecan) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive cisplatin IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Biological: bevacizumab; Drug: cisplatin; Procedure: computed tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving irinotecan and cisplatin together with bevacizumab works in treating patients with unresectable or metastatic gastric (stomach) or gastroesophageal junction adenocarcinoma (cancer). Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Giving chemotherapy together with a monoclonal antibody may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of irinotecan, cisplatin, and bevacizumab, in terms of time to progression, in patients with unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma.

SECONDARY OBJECTIVES:

I. Determine other measures of efficacy, including response rate and median and 1-year survival, in patients treated with this regimen.

II. Determine the toxicity of this regimen in these patients. III. Correlate CT perfusion imaging results with the efficacy of this regimen, in terms of time to progression, objective response, and survival, in these patients.

IV. Determine the feasibility of serial serum proteomic assays in predicting response to therapy, in terms of time to progression, objective response, and survival, in patients treated with this regimen.

V. To bank paraffin stored tumor biopsy material for future planned immunohistochemistry studies to correlate with sensitivity to bevacizumab based combination chemotherapy.

OUTLINE: This is an open-label, non-randomized, multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive cisplatin IV over 30 minutes followed by irinotecan IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric or gastroesophageal junction (GEJ) adenocarcinoma

  * Metastatic or unresectable disease
  * Siewert's classification I, II, or III
* No ulcerated, non-healing tumors or tumors that have developed a malignant fistula
* No esophageal tumors
* No known or active brain metastases
* Performance status - Karnofsky 60-100%
* Performance status - ECOG 0-2
* Neutrophil count >= 1,500/mm^3
* Platelet count >= 75,000/mm^3
* No bleeding diathesis or coagulopathy
* Bilirubin =< 1.5 mg/dL
* AST and ALT =< 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* PT (INR) =< 1.5
* PTT =< 3 seconds above ULN
* Creatinine =< 1.5 mg/dL
* Proteinuria < 1+
* Protein < 500 mg/24-hour urine collection
* No acute ischemia or significant conduction abnormality by EKG
* No clinically significant cardiovascular disease
* No uncontrolled hypertension (blood pressure > 160/90 mm Hg on medication)
* No myocardial infarction within the past 6 months
* No unstable angina within the past 6 months
* No transient ischemic attack within the past 6 months
* No cerebrovascular accident within the past 6 months
* No other arterial thromboembolic event within the past 6 months
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac dysrhythmia requiring medication
* No peripheral vascular disease (grade II or greater)
* No history of stroke
* No CNS disease within the past 5 years (e.g., uncontrolled seizures)
* No other concurrent uncontrolled illness
* No ongoing or active infection requiring parental antibiotics on Day 0 of study
* No serious, non-healing wound
* No serious wound healing by secondary intention
* No ulcer
* No bone fracture
* No psychiatric illness or social situation that would preclude study compliance
* No significant traumatic injury within the past 28 days
* No other neoplastic disease within the past 3 years except basal cell skin cancer, carcinoma in situ of the cervix, or nonmetastatic prostate cancer
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No other medical condition that would preclude study participation
* Not pregnant or nursing

  * No nursing during and for 4 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study participation
* More than 8 weeks since prior immunotherapy and recovered
* No other concurrent biologic or immunologic agents
* No other concurrent bevacizumab
* No prior chemotherapy for metastatic disease
* No prior cisplatin or irinotecan
* Prior neoadjuvant and/or adjuvant chemotherapy or chemoradiotherapy allowed
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* More than 3 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior fine needle aspirations or core biopsies
* No concurrent major surgery
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent chronic daily aspirin (> 325 mg/day)
* No concurrent nonsteroidal anti-inflammatory medications that would inhibit platelet function at doses used to treat chronic inflammatory diseases
* Full-dose anticoagulants allowed, provided the following criteria are met:

  * INR in range (i.e., 2-3) while on a stable dose of warfarin or low molecular weight heparin
  * No active bleeding or pathologic condition that would confer a high risk of bleeding (e.g., tumor involving major blood vessels or known varices)
* No concurrent thrombolytic agents
* No concurrent vitamins, antioxidants, herbal preparations, or supplements

  * Single tablet multivitamin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to progression, evaluated using RECIST | Up to 1 year
  Kaplan-Meier estimates will be used.

SECONDARY OUTCOMES:
Overall response rate, evaluated using RECIST | Up to 1 year
  95% exact binomial confidence intervals will be used to describe the distribution.
Complete response rate, evaluated using RECIST | Up to 1 year
  95% exact binomial confidence intervals will be used to describe the distribution.
Duration of response, evaluated using RECIST | From the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 1 year
Survival | Up to 1 year
  Kaplan-Meier estimates will be used.
Incidence of toxicity, evaluated using CTCAE version 3.0 | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States